CLINICAL TRIAL: NCT02091427
Title: Circadian Variation of Cardiac Troponin
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC 12-2-074
Record Dates: First submitted 2014-03-18; First posted 2014-03-19 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Individuals

SUMMARY:
Acute myocardial infarction (AMI) is defined by an increase and/or decrease in the concentration of cardiac troponin, with at least one value above the 99th percentile value of the reference population together with evidence of ischemia. An objective tool to determine the magnitude of the cardiac troponin change is the use of reference change values (RCV). The basis for this tool is that, for a change to be significant, the difference in serial results must be greater than the inherent variation in two test results. The inherent variation of a laboratory test result is composed of analytical and within-subject biological variation. An important requirement to use RCVs is that the concentrations of cardiac troponins fluctuate randomly around a homeostatic set point in cardio-healthy individuals. Verification of this important condition has never been performed, and violation of this condition would preclude the use of RCV's in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with no evidence of active cardiovascular disease

Exclusion Criteria:

* History of acute myocardial infarction in the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with no evidence of active cardiovascular disease
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
cardiac troponins | measured every hour, total time 25h (08:30 day 1, till 09:30 day 2)

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Derived] Alaour B, Kaier TE, Hasselbalch RB, van Doorn W, Meex S, Marber M. Direct Comparison of the Circadian Rhythm of Cardiac Myosin-Binding Protein C (cMyC) and Cardiac Troponin. J Appl Lab Med. 2023 Jul 5;8(4):831-834. doi: 10.1093/jalm/jfad025. No abstract available. PMID 37226050
- [Derived] Breidthardt T, van Doorn WPTM, van der Linden N, Diebold M, Wussler D, Danier I, Zimmermann T, Shrestha S, Kozhuharov N, Belkin M, Porta C, Strebel I, Michou E, Gualandro DM, Nowak A, Meex SJR, Mueller C. Diurnal Variations in Natriuretic Peptide Levels: Clinical Implications for the Diagnosis of Acute Heart Failure. Circ Heart Fail. 2022 Jun;15(6):e009165. doi: 10.1161/CIRCHEARTFAILURE.121.009165. Epub 2022 Jun 7. PMID 35670217
- [Derived] Klinkenberg LJ, Wildi K, van der Linden N, Kouw IW, Niens M, Twerenbold R, Rubini Gimenez M, Puelacher C, Daniel Neuhaus J, Hillinger P, Nestelberger T, Boeddinghaus J, Grimm K, Sabti Z, Bons JA, van Suijlen JD, Tan FE, Ten Kate J, Bekers O, van Loon LJ, van Dieijen-Visser MP, Mueller C, Meex SJ. Diurnal Rhythm of Cardiac Troponin: Consequences for the Diagnosis of Acute Myocardial Infarction. Clin Chem. 2016 Dec;62(12):1602-1611. doi: 10.1373/clinchem.2016.257485. Epub 2016 Oct 5. PMID 27707754